CLINICAL TRIAL: NCT01751867
Title: An Open-label, Multi-center, Phase IIIb Study for Decitabine in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: An Effectiveness and Safety Study of Decitabine in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017443; DACOGENMYE-3002 (Other: Xian-Janssen Pharmaceutical Ltd)
Record Dates: First submitted 2012-07-25; First posted 2012-12-18 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Dacogen; Oncology; Decitabine; Bone marrow disorders
MeSH Terms: conditions — Myelodysplastic Syndromes; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-Day Dose schedule (Experimental): Decitabine will be administered at a dose of 15 mg/m2 as a continuous intravenous infusion within a 3 hour period, repeated every 8 hours for 3 consecutive days. Cycles will be repeated every 6 weeks.
  Interventions: Drug: Decitabine at 15 mg/m2
- 5-Day Dose schedule (Experimental): Decitabine will be administered at a dose of 20 mg/m2 as a intravenous infusion within 1 hour, once daily for 5 consecutive days. Cycles will be repeated every 4 weeks.
  Interventions: Drug: Decitabine at 20 mg/m2

INTERVENTIONS:
Drug: Decitabine at 15 mg/m2 — Decitabine will be given at a dose of 15 mg/m2 as a continuous intravenous infusion within a 3-hour intravenous infusion, repeated every 8 hours for 3 consecutive days.The total dose per day is 45 mg/m2; The total dose per course is 135 mg/m2. Cycles will be repeated every 6 weeks.
  Arms: 3-Day Dose schedule
Drug: Decitabine at 20 mg/m2 — Decitabine will be given at a dose of 20 mg/m2 as 1-hour IV infusion once daily on Days 1 through 5, of a 4-week treatment cycle.
  Arms: 5-Day Dose schedule

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of decitabine in the treatment of myelodysplastic syndrome (name of a group of conditions that occur when the blood-forming cells in the bone marrow are damaged) in Chinese patients.

DETAILED DESCRIPTION:
This is a prospective (look forward using periodic observations collected predominantly following patient enrollment), open-label (all people involved in the study know the identity of the assigned drug), Phase IIIb study to evaluate the efficacy and safety of decitabine in the treatment of myelodysplastic syndrome (MDS). Patients are randomized (study drug assigned by chance) in 1:1 ratio to receive treatment with decitabine either 3-day or 5-day course of therapy. When a minimum of 30 patients are reached for 3-day course of therapy, the rest of the patients will all be enrolled into 5-day course of therapy. Each patient in the study treated for a minimum of 4 cycles; however, a complete or partial response may take longer than 4 cycles. The entire study duration for each patient will be approximately two years. Safety will be evaluated for each patient by monitoring of adverse events, physical examinations, vital signs measurements, electrocardiogram, hematology and clinical chemistry testing.

ELIGIBILITY:
Inclusion Criteria:

* Must have diagnosed with Myelodysplastic Syndrome (MDS) denovo (previously not present) or secondary as per the classification of French-American-British (FAB) and International Prognostic Scoring System (IPSS) greater than or eaul to 0.5 as determined by complete blood count (CBC), bone marrow assessment and bone marrow cytogenetics
* Must have an Eastern Oncology Cooperative Group (ECOG) performance status of 0-2
* Must have adequate hepatic and renal function as measured by the aspartate transaminase (AST), alanine transaminase (ALT), total bilirubin and serum creatinine, respectively
* Must have recovered from all toxic effects of prior therapy and not received any chemotherapy for a minimum of 4 weeks (6 weeks if the patient has been treated with a nitrosoureas) prior to the first dose of study drug - Woman must be postmenopausal, or surgically sterile, or abstinent, or, if sexually active, be practicing an effective method of birth control (eg, oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization)

Exclusion Criteria:

* Must not have a diagnosis of acute myeloid leukemia (greater than 30% bone marrow blasts) - Must not have received radiotherapy within 14 days before the first dose of study drug - Must not have any other prior cancer, other than superficial bladder cancer, basal cell skin and cervical cancer - Must not have associated autoimmune hemolytic anemia or immune thrombocytopenia and inaspirable bone marrow - Must not have a mental illness or any other condition (eg, uncontrolled cardiac or pulmonary disease, diabetes), that could prevent full cooperation with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (8):
- China (8):
  - Beijing
  - Chengdu
  - Guangdong
  - Hangzhou
  - Nanjing
  - Shanghai
  - Suzhou
  - Tianjin

REFERENCES:
- [Derived] Wu D, Du X, Jin J, Xiao Z, Shen Z, Shao Z, Li X, Huang X, Liu T, Yu L, Li J, Chen B, He G, Cai Z, Liang H, Li J, Ruan C. Decitabine for Treatment of Myelodysplastic Syndromes in Chinese Patients: An Open-Label, Phase-3b Study. Adv Ther. 2015 Nov;32(11):1140-59. doi: 10.1007/s12325-015-0263-8. Epub 2015 Nov 14. PMID 26568466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 12 centers in China.
Groups:
- 3-Day Posology: Decitabine 15 milligram per meter^2 (mg/m^2) administered by continuous intravenous infusion over a 3-hour period, repeated every 8 hours for 3 consecutive days. Cycles repeated every 6 weeks.
- 5-Day Posology: Decitabine 20 mg/m^2 administered by a 1-hour intravenous infusion once daily, on Days 1 through 5. Cycles repeated every 4 weeks.
Period: Overall Study
Arm/Group | 3-Day Posology | 5-Day Posology
Started | 36 | 99
Treated | 34 | 98
Completed | 0 | 0
Not Completed | 36 | 99
Not completed — Completed treatment,dropped in follow-up | 4 | 8
Not completed — Diease Progression | 4 | 18
Not completed — Adverse Event | 8 | 15
Not completed — Poor Compliance | 0 | 5
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 4 | 7
Not completed — Protocol Violation | 0 | 2
Not completed — Death | 0 | 5
Not completed — Other | 11 | 37
Not completed — Randomized but not treated. | 2 | 1

BASELINE CHARACTERISTICS:
Population: Randomized analysis set included all randomized participants, regardless of whether having received any treatment, or whether having any post-baseline efficacy data.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3-Day Posology | 5-Day Posology | Total
Number analyzed (Participants) | 36 | 99 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (16.04) | 51.6 (14.78) | 51.0 (15.11)
Age, Customized [Number; unit: Participants]
  18-60 Years (Y) (including 18 Y, excluding 60 Y) | 25 | 69 | 94
  Greater than or equal to (>=) 60 Y | 11 | 30 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 34 | 56
  Male | 14 | 65 | 79

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR): Number of Participants Who Achieved Either Complete Remission (CR), Partial Remission (PR), or Marrow Complete Remission (mCR) - International Working Group (IWG) 2006 Response Criteria
Description: IWG 2006 response criteria - CR: bone marrow evaluation shows less than or equal to (<=) 5% blasts; normal maturation of all cells lines (mCR), peripheral blood evaluation shows hemoglobin >= 11 gram per deciliter (g/dL), neutrophils >= 1000/mL, platelets >= 100,000/mL, 0% blasts; PR: Same as CR, except blasts decrease by >=50%, still greater than 5% in bone marrow.
Time Frame: From the date of first dose until 30 to 42 days after the last dose of the 2 years treatment period, or at time of discontinuation
Population: Intent-to-treat (ITT) population: Participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | 3-Day Posology | 5-Day Posology
Number analyzed (Participants) | 34 | 98
Participants | 10 [12.9 to 44.4] | 25 [13.9 to 31.2]
Statistical Analysis 1: Comparison: 3-Day Posology; Null Hypothesis: threshold for statistical significance = 10%; Test type: Superiority or Other; p = 0.003, Exact binomial proportion test; ORR % = 29.4, 95% CI 2-sided [15.1 to 47.5] — ORR % = Number of participants who achieved response divided by total ITT participants
Statistical Analysis 2: Comparison: 5-Day Posology; Null Hypothesis: threshold for statistical significance = 10%; Test type: Superiority or Other; p < 0.001, Exact binomial proportion test; ORR % = 25.5, 95% CI 2-sided [17.2 to 35.3]

2. Secondary Outcome: Hematological Improvement Rate: Number of Participants Who Achieved Complete Remission (CR), Partial Remission (PR) and Hematologic Improvement (HI) - International Working Group (IWG) 2006 Response Criteria
Description: IWG 2006 response criteria - CR: bone marrow evaluation shows <= 5% blasts; normal maturation of all cells lines (mCR), peripheral blood evaluation shows hemoglobin >= 11 g/dL, neutrophils >= 1000/mL, platelets >= 100,000/mL, 0% blasts; PR: Same as CR, except blasts decrease by >= 50%, still greater than 5% in bone marrow; HI: hemoglobin increase of >= 1.5 g/dL, platelet increase of >= 30,000/mL (starting with > 20,000/mL), neutrophils increase of >= 100% and > 500/μL.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population- Participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | 3-Day Posology | 5-Day Posology
Number analyzed (Participants) | 34 | 98
Participants | 16 | 47

3. Secondary Outcome: Cytogenetic Response Rate: Percentage of Participants Who Achieved Cytogenetic Response (Complete+Partial) by Status of Clinical Overall Response - International Working Group (IWG) 2006 Response Criteria
Description: As per IWG 2006 response criteria - Complete cytogenetic response: disappearance of the chromosomal abnormality without appearance of new ones; Partial cytogenetic response: At least 50% reduction of the chromosomal abnormality. Status of Clinical response - complete remission (CR); marrow CR (mCR); partial remission (PR).
Time Frame: as for outcome 1
Population: Participants who had baseline cytogenetic abnormality and had at least one post baseline cytogenetic assessments during study.
Measure: Number; unit: Percentage of Participants
Arm/Group | 3-Day Posology | 5-Day Posology
Number analyzed (Participants) | 6 | 24
Percentage of Participants
  Overall (n=6, 24) | 66.7 | 66.7
  CR+mCR+PR (n=3, 13) | 100.0 | 84.6
  CR (n=2, 3) | 100.0 | 66.7
  mCR (n=1, 10) | 100.0 | 90.0

4. Secondary Outcome: Transfusion Independence: Number of Participants Who Were Transfusion Independent
Description: A participant was considered to be transfusion independent, if the participant had no transfusions of Red Blood Cells (RBCs) or platelets for 8 consecutive weeks or more.
Time Frame: Baseline; up to 2 years
Population: Intent-to-treat (ITT) population: Participants who received at least one dose of study drug. Here, 'n' is the number of participants analyzed at specified time point.
Measure: Number; unit: Participants
Arm/Group | 3-Day Posology | 5-Day Posology
Number analyzed (Participants) | 34 | 98
Participants
  Baseline (Before First Dose) (n=34, 98) | 7 | 37
  Treatment Phase (n=34, 97) | 18 | 47

5. Secondary Outcome: Mean Percentage of Duration of Hospitalization (Relative to Days on Study Treatment)
Description: Duration of hospitalization was calculated as, total number of days a participant stayed in hospital during study treatment divided by the study treatment duration
Time Frame: Up to 2 years
Population: Intent-to-treat (ITT) population: Participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage of total days
Arm/Group | 3-Day Posology | 5-Day Posology
Number analyzed (Participants) | 34 | 98
Percentage of total days | 59.6 (34.20) | 59.2 (34.17)

6. Secondary Outcome: Overall Survival Rate: Percentage of Participants Who Survived During 6 Months and 12 Months of Treatment.
Time Frame: From the date of dosing until death or lost to follow-up for up to 2.5 years after last patient was enrolled
Population: Intent-to-treat (ITT) population- Participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 3-Day Posology | 5-Day Posology
Number analyzed (Participants) | 34 | 98
Percentage of participants
  6-month survival rate | 91.1 [74.8 to 97.0] | 84.7 [75.9 to 90.5]
  12-month survival rate | 75.9 [57.5 to 87.2] | 65.9 [55.5 to 74.4]

7. Secondary Outcome: Mean Change From Baseline to End of Treatment in Scores of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ C-30) Physical Functioning Scale
Description: EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients. It is composed of 30 items, multi-item measure (28 items) and 2 single-item measures. For the multiple item measure, 4-point scale is used and the score for each item range from "1 = not at all" to "4 = very much". Higher scores indicate worsening. The 2 single-item measure involves question about the overall health and overall quality of life which will be rated on a 7-point scale ranging from "1 = very poor" to "7 = excellent". Lower scores indicate worsening. Scores are averaged, and transformed to 0-100 scale; higher score=better level of physical functioning.
Time Frame: Baseline to end of treatment (approximately up to 2 years)
Population: Intent-to-treat (ITT) population- Participants who received at least one dose of study drug. The missing data was imputed by the Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 3-Day Posology | 5-Day Posology
Number analyzed (Participants) | 34 | 98
Scores on a scale | -5.5 (29.48) | -9.1 (26.34)

ADVERSE EVENTS:
Time Frame: From the date of informed consent signed until 30 days after last dose of study medication
Description: Safety analysis set included all participants who received at least 1 dose of study medication. Participants were analyzed according to the actual treatment received.
Arm/Group | 3-Day Posology | 5-Day Posology
Serious Adverse Events (participants affected / at risk) | 8/34 | 26/98
Other Adverse Events (participants affected / at risk) | 33/34 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3-Day Posology (N=34) | 5-Day Posology (N=98)
Pneumonia (Infections and infestations) | 1 (1) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 5 (7)
Lung infection (Infections and infestations) | 1 (1) | 4 (4)
Septic Shock (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Malignant tumour excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3-Day Posology (N=34) | 5-Day Posology (N=98)
White blood cell count decreased (Investigations) | 26 | 69
Platelet count decreased (Investigations) | 24 | 60
Neutrophil count decreased (Investigations) | 21 | 52
Haemoglobin decreased (Investigations) | 16 | 48
Alanine aminotransferase increased (Investigations) | 9 | 19
Blood albumin decreased (Investigations) | 5 | 9
Aspartate aminotransferase increased (Investigations) | 3 | 11
Blood bilirubin increased (Investigations) | 2 | 7
Blood creatinine increased (Investigations) | 1 | 6
Pyrexia (General disorders) | 22 | 54
Asthenia (General disorders) | 5 | 16
Constipation (Gastrointestinal disorders) | 6 | 15
Diarrhoea (Gastrointestinal disorders) | 6 | 16
Abdominal distension (Gastrointestinal disorders) | 6 | 10
Mouth ulceration (Gastrointestinal disorders) | 10 | 14
Abdominal discomfort (Gastrointestinal disorders) | 4 | 9
Nausea (Gastrointestinal disorders) | 0 | 10
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Vomiting (Gastrointestinal disorders) | 3 | 5
Gingival swelling (Gastrointestinal disorders) | 3 | 7
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Proctalgia (Gastrointestinal disorders) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 10 | 32
Lung infection (Infections and infestations) | 8 | 23
Infection (Infections and infestations) | 2 | 5
Pneumonia (Infections and infestations) | 7 | 8
Nasopharyngitis (Infections and infestations) | 3 | 3
Skin infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 3 | 2
Gingival infection (Infections and infestations) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 17
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 19
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 14
Decreased appetite (Metabolism and nutrition disorders) | 1 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 3 | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 6
Dizziness (Nervous system disorders) | 4 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 7
Insomnia (Psychiatric disorders) | 3 | 4
Conjunctival hyperaemia (Eye disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 1 | 7
Haematuria (Renal and urinary disorders) | 2 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 3
Palpitations (Cardiac disorders) | 0 | 6
Gingival bleeding (Gastrointestinal disorders) | 1 | 5
Gingival pain (Gastrointestinal disorders) | 2 | 2
Tongue ulceration (Gastrointestinal disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 10
Chest discomfort (General disorders) | 0 | 5
Chest pain (General disorders) | 0 | 5
Liver disorder (Hepatobiliary disorders) | 7 | 6
Anal infection (Infections and infestations) | 3 | 0
Blood potassium decreased (Investigations) | 1 | 5
Blood urea increased (Investigations) | 0 | 5
Transaminases increased (Investigations) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days